CLINICAL TRIAL: NCT00240903
Title: Revaccination of Healthy Subjects With Intramuscular Inactivated Subunit Influenza A/Vietnam/1203/2004 (H5N1) Vaccine Representing a Drifted Variant
Brief Title: Revaccination With Subunit Influenza A/Vietnam/1203/2004 (H5N1) Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-0043
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2007-03

CONDITIONS: Influenza
Keywords: revaccination, vaccination, influenza, H5N1 vaccine
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Influenza A/Vietnam/1203/2004 (H5N1; sanofi pasteur)

SUMMARY:
The purpose of this study is to determine whether having received an H5 vaccine in the past primes the immune system to respond rapidly to another dose of H5 vaccine. One hundred seventeen participants in a previous vaccine study (involving the A/Hong/Kong/97 virus) during the fall of 1998 at the University of Rochester will be eligible to enroll in this study. Participation in this study will up to 64 days and will involve donation of small samples of blood 7, 28, and 56 days after vaccination.

DETAILED DESCRIPTION:
This is an open label, phase I evaluation of a single dose of an investigational inactivated, subunit influenza A/Vietnam/1203/2004 (H5N1) vaccine in subjects who were previously vaccinated with a vaccine made from an antigenically distinct variant of H5N1. The study is designed to determine whether immunization with an antigenic variant can prime for responses to a single dose of vaccine representing the current pandemic threat. The primary objective is to determine the ability of a priming dose of rec H5 HA 1997 vaccine administered 7 years previously to result in booster responses to an inactivated subunit influenza A/Vietnam/1203/2004 (H5N1) vaccine. The secondary objectives are to 1) determine the safety of a booster dose of intramuscular inactivated subunit influenza A/Vietnam/1203/2004 (H5N1) vaccine in healthy adults, previously vaccinated with rec H5 HA 1997 vaccine and 2) evaluate the relationship between priming, levels of antigen-specific memory B and T cells , and the response to reactivation. The study will be performed at a single site, and will enroll as many previously vaccinated subjects as are available and eligible, up to a maximum of 117. Subjects will receive a single intramuscular dose of 90 mcg of the inactivated subunit influenza A/Vietnam/1203/2004 (H5N1) vaccine. Blood for assessment of antibody responses will be obtained before and at time points after vaccination. Subjects participating in the optional sub study will also have blood obtained for enumeration of memory B and T cells. Subjects will be followed for solicited adverse events for 7 days by memory aids and for 56 days for unsolicited adverse events. This study is linked to DMID protocol 08-0059.

ELIGIBILITY:
Inclusion Criteria:

1. Participant in the previous study of the rec H5 HA 1997 vaccine.
2. Male or non-pregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 65 years.
3. Females of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier method, abstinence, Depo-Provera, Norplant, oral contraceptives, contraceptive patches or other licensed, effective methods) for the entire study period.
4. In good health, as determined by medical history and a targeted physical examination, if necessary.
5. Able to understand and comply with planned study procedures.
6. Able to provide informed consent and be available for all study visits.

Exclusion Criteria:

1. Has participated in DMID 04-063 Study.
2. Has a known allergy to eggs, other components of the vaccine or latex.
3. Has a positive urine pregnancy test at screening or prior to vaccination (if female), is lactating, or has the intention to become pregnant within 3 months of enrollment in this study.
4. Is undergoing immunosuppression as a result of an underlying illness or treatment.
5. Has an active neoplastic disease or a history of any hematologic malignancy.
6. Is using oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
7. Has a history of receiving immunoglobulin or other blood products within the 3 months prior to enrollment in this study.
8. Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
9. Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
10. Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
11. Has an acute illness, including an oral temperature greater than 100.0 degrees F within one week of vaccination.
12. Received an experimental vaccine or medication within 1 month prior to enrollment in this study, or expects to receive an experimental vaccine, medication, or blood product during the 6 to 7-month study period.
13. Has a history of alcohol abuse or drug abuse (including chronic pain medication) in the last 5 years.
14. Has any condition that would, in the opinion of the site principal investigator, place the volunteer at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Result] Goji NA, Nolan C, Hill H, Wolff M, Noah DL, Williams TB, Rowe T, Treanor JJ. Immune responses of healthy subjects to a single dose of intramuscular inactivated influenza A/Vietnam/1203/2004 (H5N1) vaccine after priming with an antigenic variant. J Infect Dis. 2008 Sep 1;198(5):635-41. doi: 10.1086/590916. PMID 18694338